CLINICAL TRIAL: NCT05328557
Title: Phase Ia, Randomized Double-Blinded, Placebo-Controlled Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered CUG252 Following a Single Dose Administration in Normal Health Volunteers.
Brief Title: A Phase Ia Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered CUG252 in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cugene Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUG252-P101
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CUG252 (Experimental): Participants will be randomized in a 3:1 ratio to CUG252 or placebo. CUG252 or placebo will be administered at a single ascending dose in healthy volunteers.
  Interventions: Drug: CUG252
- Placebo (Placebo Comparator): Participants will be randomized in a 3:1 ratio to CUG252 or placebo. CUG252 or placebo will be administered at a single ascending dose in healthy volunteers.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CUG252 — CUG252 will be administered by subcutaneous (SC) injection
  Arms: CUG252
Drug: Placebo — Placebo will be administered by subcutaneous (SC) injection
  Arms: Placebo

SUMMARY:
The intent of this study is to evaluate the safety and tolerability of single escalating subcutaneous doses of CUG252 in healthy adult subjects.

DETAILED DESCRIPTION:
This is a Phase Ia study of CUG252, comprising a randomized, double-blind, placebo-controlled, single ascending dose in healthy adult subjects.

ELIGIBILITY:
For healthy subject cohorts,

Inclusion Criteria:

* Non-smoking adult healthy male and female, aged 18 to 65 years (inclusive), at the time of consent with a body mass index (BMI) between 18.0 and 32.0 kg/m2 (inclusive), at Screening.
* Healthy as determined by medical history, physical examination, vital signs, clinical laboratory safety tests, ECG, and chest X-ray

Exclusion Criteria:

* Active bacterial, viral, fungal infection or known inflammatory process, infection or antibiotic treatment
* Laboratory test results outside the local reference range and deemed clinically significant
* History of chronic medications, immunosuppressant or steroids
* History of malignant neoplasm
* History of relevant atopy
* History of hypersensitivity to biologic agents or any of the excipients in the formulation.
* Excessive xanthine consumption
* History of drug or alcohol addiction or dependence within 1 year
* Positive of a tuberculosis test or a history of tuberculosis
* Abnormal blood pressure and/or ECG parameters
* Any prescribed medications within 28 days or nonprescription drugs within 7 days
* Previously received aldesleukin or any other IL-2 derivative

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with Treatment Emergent Adverse Events | Up to 10 weeks
  To evaluate the safety and tolerability of subcutaneous injections of CUG252 in healthy subjects.

SECONDARY OUTCOMES:
Pharmacokinetics profile of CUG252 (AUC) | Up to 10 weeks
  To assess the Area under the plasma concentration versus time curve (AUC)
Pharmacokinetics profile of CUG252 (Cmax) | Up to 10 weeks
  To assess the maximum plasma concentration (Cmax)
Pharmacokinetics profile of CUG252 (Tmax) | Up to 10 weeks
  To assess the time of maximum concentration (Tmax)
Pharmacokinetics profile of CUG252 (t1/2) | Up to 10 weeks
  To assess the half-life (t1/2)
Immunogenicity of CUG252 | Up to 10 weeks
  To measure the serum concentration of antibodies against CUG252
Change in the number and percentages of immune cells | Up to 10 weeks
  To assess the effect of CUG252 on immuno-pharmacodynamic endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Kankam, MD, PhD, Principal Investigator — Altasciences Company Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States